CLINICAL TRIAL: NCT02211716
Title: Physician-Initiated PMCF Trial Investigating the BeGraft Peripheral Stent Graft System for the Treatment of Iliac Lesions
Brief Title: Physician-Initiated Trial Investigating the BeGraft Peripheral Stent Graft System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-131216
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BeGraft (Experimental): Patient's treated with the BeGraft PMCF Stent Graft System from Bentley Innomed for the treatment of iliac lesions.
  Interventions: Device: BeGraft Peripheral Stent Graft System

INTERVENTIONS:
Device: BeGraft Peripheral Stent Graft System

SUMMARY:
The objective of this clinical investigation is to evaluate, in a controlled setting, the long-term (up to 12 months) safety and efficacy of the BeGraft Peripheral Stent Graft System (Bentley InnoMed) in clincial settings post CE-certification when used according to the indications of the IFU.

DETAILED DESCRIPTION:
Endovascular techniques are well accepted in the treatment of iliac occlusive disease. It is shown that in the iliac artery especially stenoses and short occlusions respond well to percutaneous transluminal angioplasty (PTA) with our without stenting. Although hard data are lacking, with the technical developments and the introduction of new stent types, more complex lesions have been treated with endovascular procedures. Although stents are often used to improve the outcome of PTA, there is no general consensus whether stenting is mandatory for chronic iliac arterial occlusion. The more, if we use stents, it is still unclear if we should implant bare self-expandable stents, bare balloon-expandable stents or covered stents. On one hand, the randomized controlled Dutch Iliac Stenting trial failed in demonstrating superiority of primary stenting over PTA with additional stenting in short lesions. On the other hand, while several papers advocate bare stenting, other trials conclude better results with covered stents.

The Trans-Atlantic Inter-Society Consensus (TASC) working group has published in 2000 their recommendations for the management of peripheral arterial disease. In order to better reflect the developments in technology and techniques, the TASC working group has revised and updated their recommendations in the TASC-II document in 2007.

The treatment recommendations between surgical or percutaneous intervention they propose involve all peripheral arterial beds and are based upon several factors such as availability of expertise in the percutaneous or conventional vascular surgical techniques, the patient's preference and most importantly on the lesion's morphology. TASC classifies all lesions in the different beds into types A to D. In general, endovascular therapy is the treatment of choice for TASC A & B-lesions and surgery is preferred for good-risk patients with TASC C lesions and all TASC D lesions.

For aorto-iliac lesions, the TASC-II classification is as follows:

Type A lesions

1. Unilateral or bilateral stenoses of the Common Iliac Artery (CIA).
2. Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery (EIA).

Type B lesions

1. Short (≤3 cm) stenosis of infrarenal aorta.
2. Unilateral CIA occlusion.
3. Single or multiple stenosis totaling 3-10 cm involving the EIA not extending into the Common Femoral Artery (CFA)
4. Unilateral EIA occlusion not involving the origins of Internal Iliac Artery (IIA) or CFA Type C lesions

1. Bilateral CIA occlusions 2. Bilateral EIA stenoses 3-10 cm long not extending into the CFA 3. Unilateral EIA stenosis extending into the CFA 4. Unilateral EIA occlusion that involves the origins of IIA and/or CFA 5. Heavily calcified unilateral EIA occlusion with or without involvement of origins of IIA and/or CFA Type D lesions

1. Infra-renal aortoiliac occlusion
2. Diffuse disease involving the aorta and both iliac arteries requiring treatment
3. Diffuse multiple stenoses involving the unilateral CIA, EIA and CFA
4. Unilateral occlusions of both CIA and EIA
5. Bilateral occlusions of EIA
6. Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery

The TASC working group has based their recommendations on the literature available to date and are generally considered as the guidelines to be followed. Nevertheless it should be stated that it is feasible to treat with good technical success and sustained durability TASC type C and D lesions in an endovascular way.

Recent publications finally start to show the excellent durability of iliac stenting in the daily practice. Park et al, described their long term (up to 10 years) experience in their total cohort of iliac patients (TASC type A-D lesions) and presented impressive primary patency rates of 87%, 83%, 61% and 49% at respectively 3, 5, 7 and 10 years after the index intervention. De Roeck et al. published their results after stenting of different types of iliac occlusions (TASC type B-D), and showed primary patency rates of 94%, 89% and 77% after respectively 1, 3 and 5 years follow up. They could also show that in their cohort of patients with complex aorto-iliac lesions, stent-failures can always be endovascularly rescued. They showed secondary patency rates of 100% after 1 year and 94% after both 3 and 5 years. Bosiers et al. concluded in their BRAVISSIMO trial primary patency rates at 12 months for the TASC A, B, C and D lesions of respectively 94.0%, 96.5%, 91.3% and 90.2%. Leville et al. questioned after the presentation of their outcome with stenting iliac occlusion (primary patency rate of 76% and secondary patency rate of 90% after 3 years), whether the endovascular treatment for iliac occlusive disease should be extended to Type C and D lesions. Leville came to this conclusion as they could not detect any significant differences in outcome for both primary and secondary patency rates stratifying for the TASC classifications. They summarized the treatment of iliac artery occlusion can be accomplished via endovascular means with little morbidity and acceptable patency rates. The COBEST trial demonstrates that covered and bare-metal stents produce similar and acceptable results for TASC B lesions. However, covered stents perform better for TASC C and D lesions than bare stents in longer-term patency and clinical outcome. Sabri et al. concluded that the use of covered balloon-expandable kissing stents for atherosclerotic aortic bifurcation occlusive disease provides superior patency at 2 years as compared with bare metal balloon-expandable stents. Bosiers et al. experienced that the implantation of the Advanta V12 PTFE-covered stent for iliac occlusive disease shows to be safe and feasible with excellent clinical results at 1 year in the investigated patient cohort. The TASC stratification is an important tool in allowing us to assess the extent of lesion morphology, but extensive lesions do not preclude successful endovascular treatment. They continued that the fate of the limb is dictated by the infrainguinal disease that is often present in patients with complex iliac occlusions and therefore believe that endovascular attempts should be exhausted before attempting open surgical repair of iliac occlusions because of the decreased perioperative morbidity and good mid-term durability.

ELIGIBILITY:
Inclusion Criteria

1. General Inclusion criteria

   * Corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.
   * Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
   * Patient presenting a score from 2 to 5 following Rutherford classification
   * Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
   * Patient is >18 years old
   * Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
   * Patient is eligible for treatment with the BeGraft Peripheral Stent Graft System (Bentley InnoMed)
2. Angiographic Inclusion Criteria

   * The target lesion is either a modified TASC-II class A, B, C or D lesion with one of the listed specifications:

     * Type A lesions

       * Unilateral or bilateral stenoses of the Common Iliac Artery
       * Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery
     * Type B lesions

       * Unilateral Common Iliac Artery occlusion
       * Single or multiple stenosis totaling 3-10 cm involving the External Iliac Artery not extending into the Common Femoral Artery
       * Unilateral External Iliac Artery occlusion not involving the origins of Internal Iliac Artery or Common Iliac Artery
     * Type C lesions

       * Bilateral Common Iliac Artery occlusions
       * Bilateral External Iliac Artery stenoses 3-10 cm long not extending into the Common Femoral Artery
     * Type D lesions

       * Unilateral occlusions of both Common Iliac and External Iliac Artery
       * Diffuse disease involving the aorta and both iliac arteries requiring treatment
       * Bilateral occlusions of External Iliac Artery
   * The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
   * There is angiographic evidence of a patent Common an Deep Femoral Artery

Exclusion Criteria

* PTA is technically not possible (not feasible to access the lesion or a defect with the guidewire or balloon catheter)
* Presence of an aneurysm immediately adjacent to the site of stent implantation
* Stenosis distal to the site of stent implantation
* Lesions in or adjacent to essential collateral(s)
* Lesions in locations subject to external compression
* Heavily calcified lesions resistant to PTA
* Patients with diffuse distal disease resulting in poor stent outflow
* Patients with a history of coagulation disorders
* Patients with aspirin allergy or bleeding complications and patients unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or non-responders to anticoagulant/antiplatelet therapy
* Fresh thrombus formation
* Patients with known hypersensitivity to the stent material (L605) and/or PTFE
* The target lesion is either a modified TASC-II class B or D lesion with aortic or common femoral lesion involvement:

  * Type B lesions

    * Short (≤3 cm) stenosis of infrarenal aorta
  * Type C lesions

    * Unilateral External Iliac Artery stenosis extending into the Common Femoral Artery
    * Unilateral External Iliac Artery occlusion that involves the origins of the Internal Iliac and/or Common Femoral Artery
    * Heavily calcified unilateral External Iliac Artery occlusion with or without involvement of origins of the Internal Iliac and/or Common Femoral Artery
  * Type D lesions

    * Infra-renal aortoiliac occlusion
    * Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery
    * Diffuse multiple stenoses involving the unilateral Common Iliac, External Iliac and Common Femoral Artery
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for the available stent design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months | 12 months
  Defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.4) and without Target Lesion Revascularization (TLR) within 12 months.

SECONDARY OUTCOMES:
Primary patency rate at 1- and 6-month follow-up | 1 and 6 months
  Patients that present wihout a hemodynamically significant stenosis at the target area on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.4) and without prior TLR.
Stent graft occlusion rate at pre-discharge, 1-, 6- and 12-month follow-up | 1 day post-op, 1, 6 and 12 months
  The ratio of patients where the implanted stent graft has been occluded.
Ankle Brachial Index (ABI) at 1-, 6- and 12-month follow-up | 1, 6 and 12 months
  The ABI measurement at 1, 6 and 12 months compared to the baseline ABI measurement.
Performance success rate at baseline | 1 day post-op
  Defined as a composite of:
  * successful in sealing acute perforation or rupture
  * successful in treating aneurysms and fistulae
  * restoration of blood flow
In-stent restenosis rate at 1-, 6- and 12-month follow-up | 1, 6 and 12 months
  The ratio of patients experiencing in-stent restenosis at the different follow-ups.
Freedom from Target Lesion Revascularization (TLR) at 1-, 6- and 12-months | 1, 6 and 12 months
  Defined as freedom from a repeat intervention to maintain or re-estabish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge.
Serious Adverse Avents | up to 12 months
Technical success | 1 day post-op
  Defined as the ability to achieve final residual angiographic stenosis no greater than 30%.
Amputation rate at 1-, 6- and 12-month follow-up | 1, 6 and 12 months
  Defined as any amputation above the knee.
Clinical success at 1-, 6- and 12-month follow-up | 1, 6 and 12 months
  Defined as an improvement of Rutherford classification at 1-, 6- and 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — Flanders Medical Research Program
Locations (4):
- Belgium (4):
  - OLV Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - RZ Heilig Hart Tienen, Tienen

IPD SHARING:
Plan to Share IPD: Undecided